CLINICAL TRIAL: NCT04767841
Title: The AMPK Modulator Metformin as a Novel Adjunct to Conventional Therapy in Patients With Knee Osteoarthritis: A Proof-of-Concept, Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: The AMPK Modulator Metformin as a Novel Adjunct to Conventional Therapy in Patients With Knee Osteoarthritis
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Institutional and funding constrains
Sponsor: Sadat City University (Other)
Responsible Party: Principal Investigator, Mahmoud Samy Abdallah, Principle Investigator, Sadat City University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10/2021RHU
Record Dates: First submitted 2021-02-16; First posted 2021-02-23 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Osteo Arthritis Knee
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Experimental): Metformin 1000 mg daily plus Celecoxib 200mg capsule
  Interventions: Drug: Metformin
- Placebo (Experimental): Placebo tablet daily plus Celecoxib 200mg capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin 1000mg tablet plus celecoxib 200 mg capsule
  Arms: Metformin
Drug: Placebo — Placebo tablet plus celecoxib 200 mg capsule
  Arms: Placebo

SUMMARY:
metformin alleviates drug-induced osteoarthritis (OA)-like change in mice knee joint through activating autophagy and downregulating apoptosis. Metformin exerts its protective effects against OA through the AMPKa2/ SIRT1 pathway. Metformin suppresses IL-1β-induced oxidative and osteoarthritis-like inflammatory changes by enhancing the SIRT3/PINK1/Parkin signaling pathway, thereby indicating metformin's potential in prevention and treatment of osteoarthritic joint disease.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis Patients recruited were between 30 to 60 years of age, with X-ray confirmed Kellgren-Lawrence grade13 II or III severity primary tibiofemoral OA, according to the American College of Rheumatology criteria.

Exclusion Criteria:

Those patients were excluded from the present study who:

* were of age less than 30 years or more than 60 years
* presented with active concomitant gastroduodenal disorders, hepatic and renal impairment within last 30 days prior to receiving the study drug
* were diagnosed to have any inflammatory arthritis, gout or acute trauma of the knee, hip or spine; accompanying OA of the hip of sufficient severity to interfere with the functional assessment of the knee
* had previous or ongoing treatment with oral SYSDOA (e.g., glucosamine sulphate, chondroitin sulphate, diacerein, piascledine), anti-depressants, tranquillisers, antacids or antibiotics; were having active cardiac lesion or hypertension, were pregnant females and those who were planning their pregnancy during the study
* were having a known hypersensitivity to the used medications
* have persistent diarrhoea or laxative use; severe gastrointestinal disorders, severe obesity, severe parenchymal organ disease, or anaemia (haemoglobin< 10.0 g/ dl or haematocrit < 30%).
* Patients who received oral, intramuscular, intraarticular or soft tissue injections of corticosteroids within last eight weeks before receiving the first dose of the study medication, or had undergone joint lavage and arthroscopic procedures in the previous 6 months, were also excluded.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue scale assessment of pain | week 12
  the change of Visual Analogue Scale (VAS) pain score from baseline to posttreatment

SECONDARY OUTCOMES:
WOMAC change | week 12
  the change of WOMAC Osteoarthritis Index from baseline to posttreatment
the change of Short Form 36 Questionnaire (SF-36) score from baseline to posttreatment | week 12
  The SF-36 is a generic instrument to assess health-related quality of life. It consists of 36 questions and assesses 8 dimensions: physical functioning, role physical, pain index, general health, vitality, social functioning, role emotional, and mental health index. It also provides 2 summary measures of physical and mental components. The SF-36 score ranges from 0 to 100, with higher scores indicating better health status.
Adverse drug reaction | 12 weeks
  Clinical side effects
AMPK expression | 12 weeks
  AMPK gene expression
Serum level Tumor necrosis factor- alpha (TNF-α) | 12 weeks
  Serum level Tumor necrosis factor- alpha (TNF-α)
Serum levels of IL-1β | 12 weeks
  Serum levels of IL-1β
IL-17 | 12 weeks
  Serum levels of IL-17

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF